CLINICAL TRIAL: NCT00627874
Title: A Randomised, Controlled Trial of Prevention of Juvenile-Onset Myopia in Chinese Children
Brief Title: Trial of Myopia Prevention Using +3D Lenses
Acronym: PLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Australian National University (Other)
Responsible Party: Mingguang He, Zhongshan Ophthalmic Center, ZOC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PLS2008
Record Dates: First submitted 2008-02-20; First posted 2008-03-04 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

ARMS (2):
- 1 (Experimental): wear +3D glasses for 30 minutes per day and engage in activities which require vision at more than 1m
  Interventions: Device: +3D Lenses
- 2 (No Intervention)

INTERVENTIONS:
Device: +3D Lenses — wear +3D glasses for 30 minutes per day and engage in activities which require vision at more than 1m
  Arms: 1

SUMMARY:
The purpose of this study is to assess whether a short-term imposed myopic defocus is effective in preventing the development and progression of juvenile-onset myopia in Chinese children.

DETAILED DESCRIPTION:
1. To determine if +3D lenses wearing for half an hour everyday prevents the development and progression of myopia in school children.
2. To identify ocular parameters and risk factors at baseline associated with development and progression of myopia.

ELIGIBILITY:
Inclusion Criteria:

* All children in the selected class are enrolled

Exclusion Criteria:

* Hyperopia > +2.0 D
* High myopia > -6.0 D
* Astigmatism> 1.5 D
* Anisometropia > 1.5 D
* Strabismus and amblyopia
* Any ocular, systemic, or neurodevelopmental conditions that could influence refractive development
* Chronic medication use that might affect myopia progression or visual acuity
* Already receiving other treatment for progressing myopia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Axial Length of eyes | Annual

SECONDARY OUTCOMES:
Autorefraction | Annual

CONTACTS AND LOCATIONS:
Overall Officials: Mingguang He, PhD, MD, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University